CLINICAL TRIAL: NCT00287885
Title: Phase I Study of Metronomic Daily Dosing of Docetaxel in Women With Progressive or Recurrent Gynecologic Cancer
Brief Title: Docetaxel in Treating Patients With Refractory or Recurrent Advanced Gynecologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2003LS034; UMN-WCC-35 (Other: Women's Cancer Center, University of Minnesota); 0307M50626 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Cervical Cancer; Endometrial Cancer; Fallopian Tube Cancer; Ovarian Cancer; Peritoneal Cavity Cancer; Sarcoma; Vaginal Cancer; Vulvar Cancer
Keywords: recurrent cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; stage III endometrial carcinoma; recurrent endometrial carcinoma; stage IV endometrial carcinoma; fallopian tube cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; stage III ovarian germ cell tumor; recurrent ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian epithelial cancer; recurrent uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; stage III vaginal cancer; recurrent vaginal cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; stage III vulvar cancer; recurrent vulvar cancer; stage IV vulvar cancer; ovarian sarcoma; ovarian stromal cancer; peritoneal cavity cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms; Sarcoma; Vaginal Neoplasms; Vulvar Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metronomic Docetaxel (Experimental): Docetaxel will be administered by daily injection via pre-filled syringes into the patient's accessed subcutaneous port.
  Interventions: Drug: docetaxel

INTERVENTIONS:
Drug: docetaxel — Three patients will be enrolled and dosed at each level; from dose level 1 of 2.9 mg/m^2/day up to dose level 6 of 6.4 mg/m^2/day
  Other Names: Taxotere

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Docetaxel may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving daily doses of docetaxel may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of docetaxel in treating patients with refractory or recurrent advanced gynecologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of metronomic docetaxel in patients with progressive or recurrent gynecologic cancer.

Secondary

* Determine the response rate in patients treated with this drug.
* Determine the pharmacokinetics associated with this drug in these patients.

OUTLINE: This is a dose-escalation study.

Patients receive docetaxel intravenously (IV) over 1-2 minutes daily for up to 6 months in the absence of unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of docetaxel until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed advanced, refractory gynecologic cancer.
* Patients must have received prior chemotherapy, and must have residual or recurrent disease after initial therapy or after subsequent therapy.
* Patients must have at least one site of bi-dimensional measurable disease as defined in section 9 or must have evaluable but radiographically non-measurable disease associated with CA-125 > 50 units/ml on two measurements at least one week apart. Baseline measurements and CA-125 must be obtained for all patients within four weeks before registration.
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Patients must not have received any hormonal or immunologic therapy for 2 weeks or cytotoxic chemotherapy or radiation therapy for 4 weeks (nitrosoureas and mitomycin C require 6 weeks) prior to registration.
* Patients may not have a history of prior malignancy in the past 5 years other than non-melanoma skin cancer or in situ carcinoma of the cervix.
* Patients must have documented adequate organ function within 4 weeks of registration defined as:

  * Marrow: WBC ≥ 3000/mm3, ANC ≥ 1500/mm3 , Hgb ≥ 8.0 g/dl, platelets ≥ 100,000/mm3
  * Hepatic: Total Bilirubin ≤ ULN, SGOT or SGPT and Alkaline Phosphatase must be within the range allowing for eligibility, as in the table below
  * SGOT or SGPT: Meets 1 of the following criteria:

    * Alkaline phosphatase (AP) normal AND SGOT or SGPT normal
    * AP ≤ 5 times ULN AND SGOT or SGPT normal
    * AP normal AND SGOT or SGPT ≤ 5 times ULN
    * AP ≤ 2.5 ULN AND SGOT or SGPT ≤ 1.5 times ULN
  * Renal: BUN ≤ 30 mg%, creatinine ≤ 1.5 mg%
* Age ≥ 18 years

Exclusion Criteria:

* Pregnant or lactating. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk.
* Patients of reproductive potential must use effective birth control, preferably with barrier methods.
* Prior history of myocardial infarction, congestive heart failure or significant ischemic or valvular heart disease.
* Patients with known brain metastases are not eligible.
* Peripheral neuropathy must be ≤ grade 2.
* Patients with a history of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80 must be excluded.

Patient must given written informed consent indicating the investigational nature of the treatment and its potential risks

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2004-03; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 180 Days
  Determine the maximum tolerated dose of metronomic docetaxel in patients with progressive or recurrent gynecologic cancer

SECONDARY OUTCOMES:
Response to Treatment | Up to 180 Days
  Determine the response rate in patients treated with this drug.
Pharmacokinetics | Day 1 through Day 5
  Determine the pharmacokinetics associated with this drug in these patients.

CONTACTS AND LOCATIONS:
Overall Officials: Levi S. Downs, MD, Study Chair — Masonic Cancer Center, University of Minnesota